CLINICAL TRIAL: NCT03766282
Title: Pharmacokinetics of Antibiotics, Sedative and Analgesic During Extracorporeal Membrane Oxygenation
Brief Title: Pharmacokinetics in Extracorporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, Prof., China-Japan Friendship Hospital
Other Study IDs: 2017-2-QN-15
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Extracorporeal Membrane Oxygenation; Pharmacokinetics
Keywords: Pharmacokinetics; extracorporeal membrane oxygenation
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples drawn from an existing arterial line and collect in 2-4ml tubes. Centrifuged at 3000 rpm for 10 minutes before frozen at -80℃.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Animal study: Critically ill animal on ECMO. PK data from critically ill animal on ECMO will be compared with data from controls and healthy animal on ECMO.
  Interventions: Device: ECMO
- Clinical study: To describe variation of plasma concentration of drugs in patients receiving ECMO, as compared with patients without ECMO.And develop population PK model for ECMO patients.
  Interventions: Device: ECMO

INTERVENTIONS:
Device: ECMO — Extracorporeal membrane oxygenation (ECMO) temporarily supports patients with severe cardio-respiratory failure
  Other Names: Extracorporeal membrane oxygenation

SUMMARY:
The main purpose of the present study is to investigate the risk factors that affect drug pharmacokinetic (PK) during extracorporeal membrane oxygenation (ECMO). To advance understanding of PK variance and improve the patients outcomes during ECMO.

DETAILED DESCRIPTION:
Ex vivo experiments for drug stability testing and ECMO circuits testing in animal models.PK studies in healthy animals and critically ill animal models with or without ECMO to define the PK alterations. Clinical PK studies in critically ill patients on ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing ECMO for respiratory and or cardiac dysfunction
* Clinical indication for the antibiotics
* Clinical indication for the sedatives and analgesics

Exclusion Criteria:

* No consent
* Known allergy to study drug
* Pregnancy
* Massive fluid resuscitation (>50% blood volume transfused) in the previous 8 hours.
* Therapeutic plasma exchange in the preceding 24 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing ECMO
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The median observed peak concentration(Cmax) | one-dose period
  Using liquid chromatography-mass spectrometry to evaluate the concentration of study drugs
The median observed through concentration(Cmin) | one-dose period
  Using liquid chromatography-mass spectrometry to evaluate the concentration of study drugs
Volume of distribution(Vd) | one-dose period
  PK data were analyzed with a nonlinear mixed-effect modeling approach using NONMEM version 7.2.0
Area under the plasma concentration versus time curve (AUC) | one-dose period
  PK data were analyzed with a nonlinear mixed-effect modeling approach using NONMEM version 7.2.0
Inter-compartmental clearance (Q) | one-dose period
  PK data were analyzed with a nonlinear mixed-effect modeling approach using NONMEM version 7.2.0
Clearance(CL) | one-dose period
  PK data were analyzed with a nonlinear mixed-effect modeling approach using NONMEM version 7.2.0

SECONDARY OUTCOMES:
Development of strategies for drug administration in critically ill patients receiving ECMO | one-dose period
  PK models for study drugs using a non-linear mixed effects modeling approach.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Q, Zhang Z, Liu D, Chen W, Cui G, Li P, Zhang X, Li M, Zhan Q, Wang C. Population Pharmacokinetics of Caspofungin among Extracorporeal Membrane Oxygenation Patients during the Postoperative Period of Lung Transplantation. Antimicrob Agents Chemother. 2020 Oct 20;64(11):e00687-20. doi: 10.1128/AAC.00687-20. Print 2020 Oct 20. PMID 32816724